CLINICAL TRIAL: NCT02376413
Title: Prospective Non-randomized Evaluation of Oncoplastic Breast-conserving Surgery in Non-metastatic Breast Cancer Patients
Brief Title: Oncoplastic Breast-conserving Surgery in Non-metastatic Breast Cancer Patients
Status: Withdrawn | Type: Observational
Why Stopped: Unavailable to recruit patients.
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Erwei Song, M.D., Ph.D., Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: sysubcr001
Record Dates: First submitted 2015-02-17; First posted 2015-03-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Local Recurrence of Malignant Tumor of Breast
Keywords: Morbidity; The Breast Cancer Treatment Outcome Scale; Disease free survival; Positivity cavity margin rate; Harvard/NSABP/RTOG breast cosmesis grading scale
MeSH Terms: interventions — Mastectomy, Segmental; Drug Therapy; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Traditional BCS: Breast-conserving surgery. Modified radical mastectomy.
  Interventions: Procedure: Breast surgery; Drug: Chemotherapy or endocrine therapy or Trastuzumab therapy; Radiation: Radiation therapy
- Oncoplastic-BCS: Breast-conserving surgery. Modified radical mastectomy. Oncoplastic-BCS based on surgeon preference and/or tumor location.
  * Superior pedicle mammoplasty / inverted T
  * Superior pedicle mammoplasty / V scar
  * Batwing
  * Inferior pedicle mammoplasty
  * Racquet mammoplasty/radial scar
  * vertical-scar mammoplasty
  Interventions: Procedure: Breast surgery; Drug: Chemotherapy or endocrine therapy or Trastuzumab therapy; Radiation: Radiation therapy

INTERVENTIONS:
Procedure: Breast surgery — Traditional breast-conserving surgery, oncoplastic breast-conserving surgery or modified radical mastectomy
Drug: Chemotherapy or endocrine therapy or Trastuzumab therapy
Radiation: Radiation therapy

SUMMARY:
Breast-conserving surgery (BCS) is the traditional surgical treatment for early-stage breast cancer patients. There are evidences indicating that oncoplastic-BCS (displacement technique) could improve cosmetic outcomes and/or quality of life, and has similar oncological safety as traditional BCS does. However, there are no prospective trial comparing oncoplastic-BCS vs. traditional BCS in terms of cosmetic outcomes and oncological safety. In this study, the investigators are going to address this issue by assigning patients into traditional and oncoplastic-BCS group, based on their preference.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* ECOG<=2
* Non-metastatic breast cancer patients with unilateral breast cancer confirmed by pathology.
* Operable or operable after neoadjuvant chemotherapy.
* Extensive, diffuse micro-calcifications on mammography before surgery
* No history of breast surgery or breast radiation therapy before.
* Able to follow the standard of care in adjuvant chemotherapy, radiation therapy, endocrine therapy and targeted therapy after surgery.

Exclusion Criteria:

* Multifocal/multicentric diseases noticed before surgery.
* Inflammatory breast cancer or invasive micro-papillary carcinoma of the breast confirmed by pathology before surgery.
* Tumor size > 5 cm revealed by physical examination, Ultrasound or mammography before surgery.
* Tumor size/breast size ratio >0.5 revealed by by physical examination, Ultrasound or mammography before surgery.
* Have other malignant tumors.
* Have severe co-morbidities that compromise the patients' compliance to our protocol, or endanger the patients.
* Participated in other clinical trials.
* Pathologically confirmed metastatic breast cancer, bilateral breast cancer or DCIS patients.
* Patients with any organ failure.
* Pregnancy women
* Patients who desire to have mastectomy before surgery.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-metastatic breast cancer patients received surgical treatment in Sun Yat-sen Memorial Hospital, Sun Yat-sen University. Informed consent must be obtained for all of the included patients.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Harvard/NSABP/RTOG breast cosmesis grading scale | 5 years

SECONDARY OUTCOMES:
Positivity rate of cavity margin | Intraoperatively.
Local-recurrence free survival | 5 years
Disease free survival | 5 years
Breast Cancer Treatment Outcome Scale (BCTOS) | 5 years
Morbidity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Erwei Song, M.D. Ph.D., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Fengxi Su, M.D., Study Director — Yat-sen Memorial Hospital, Sun Yat-sen University.